CLINICAL TRIAL: NCT00835848
Title: Pharmacological Postconditioning to Reduce Infarct Size Following Primary PCI in Patients With STEMI
Brief Title: Pharmacological Postconditioning to Reduce Infarct Size Following Primary PCI
Acronym: POSTCON II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Thomas Engstrom, Chief consultant, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KF 01 326257 b
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Myocardial Infarction
Keywords: ST-segment elevation myocardial infarction; Primary PCI; Postconditioning
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction | interventions — Exenatide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Exenatide (Active Comparator): 25 μg Byetta (Lilly, Exenatide) is added to 250 ml isotonic NaCl. Infusion is started immediately at 72ml/hour for 15 min, followed by 26ml/hour to be contoinued for 6 hours.
  Interventions: Drug: Exenatide
- Saline (Placebo Comparator): Isotonic saline infusion is started immediately at 72ml/hour for 15 min, followed by 26ml/hour to be contoinued for 6 hours.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Exenatide — Following arrival at the catheter laboratory informed consent is obtained and the patient randomised to placebo or exenatid treatment. 25 μg Byetta (Lilly, Exenatide) and 0.1% human albumine are added to 250 ml isotonic NaCl. Infusion is started immediately at 72ml/hour for 15 min, followed by 26ml/hour to be contoinued for 6 hours.
  Arms: Exenatide
Drug: Saline — Following arrival at the catheter laboratory informed consent is obtained and the patient randomised to placebo or exenatid treatment. 0.1% human albumine is added to 250 ml isotonic NaCl. Infusion is started immediately at 72ml/hour for 15 min, followed by 26ml/hour to be contoinued for 6 hours.
  Arms: Saline

SUMMARY:
Both pre- and postconditioning seem to protect cardiomyocytes during reperfusion therapy. Investigations both ex vivo and in vivo suggest that a gut derived hormone, Glucagon-Like-Peptide-1 (GLP-1), is able to reduce reperfusioninjury after myocardial ischemia. Results from our own laboratory have shown a marked reduction in infarct size when rat hearts in a Langendorf preparation were exposed to the GLP-1 analogue, exendin-4. The investigators want to investigate to what extent this effect can be translated to humans in the setting of acute STEMI treated with primary PCI when evalutaed by cardiac magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years of age.
* STEMI less than 12 hours from onset of pain. STEMI defined as as ST-segment elevation in 2 contiguous electrocardiographic leads of >0.1 mV in V4 - V6 or limb leads II, III and aVF, or >0.2 mV in lead V1 - V3.
* TIMI 0-1 in infarct related artery.
* Oral and written informed consent.

Exclusion Criteria:

* Multivessel disease defined by one or more stenoses >70% in diameter in the non infarct related artery.
* Previous myocardial infarction.
* Stent trombosis.
* Previous CABG.
* Less than TIMI 2 following wiring and predilatation of the infarct related artery but prior to postconditioning or placebo treatment.
* Renal insufficiency (creatinin >200).
* Pregnancy or lactation.
* Diabetic ketoacidose eller hypoglycemia (plasma glukose < 2.5 mmol/l).
* Pancreatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Infarct size by MRI | 3 months

SECONDARY OUTCOMES:
Cardiel death after 1 and 15 months. | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Engstrom, MD, PhD, DSci, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Heart Center, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Huang M, Wei R, Wang Y, Su T, Li Q, Yang X, Chen X. Protective effect of glucagon-like peptide-1 agents on reperfusion injury for acute myocardial infarction: a meta-analysis of randomized controlled trials. Ann Med. 2017 Nov;49(7):552-561. doi: 10.1080/07853890.2017.1306653. Epub 2017 Mar 31. PMID 28286967
- [Derived] Lonborg J, Kelbaek H, Vejlstrup N, Botker HE, Kim WY, Holmvang L, Jorgensen E, Helqvist S, Saunamaki K, Terkelsen CJ, Schoos MM, Kober L, Clemmensen P, Treiman M, Engstrom T. Exenatide reduces final infarct size in patients with ST-segment-elevation myocardial infarction and short-duration of ischemia. Circ Cardiovasc Interv. 2012 Apr;5(2):288-95. doi: 10.1161/CIRCINTERVENTIONS.112.968388. Epub 2012 Apr 10. PMID 22496084
- [Derived] Lonborg J, Vejlstrup N, Kelbaek H, Botker HE, Kim WY, Mathiasen AB, Jorgensen E, Helqvist S, Saunamaki K, Clemmensen P, Holmvang L, Thuesen L, Krusell LR, Jensen JS, Kober L, Treiman M, Holst JJ, Engstrom T. Exenatide reduces reperfusion injury in patients with ST-segment elevation myocardial infarction. Eur Heart J. 2012 Jun;33(12):1491-9. doi: 10.1093/eurheartj/ehr309. Epub 2011 Sep 14. PMID 21920963